CLINICAL TRIAL: NCT07220447
Title: Investigating the Feasibility and Relationship of L-Theanine in Supporting Relaxation and Mood in Cancer Patients in Surveillance
Brief Title: L-Theanine to Support Relaxation and Mood for Cancer Patients in Surveillance
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24886; NCI-2025-05686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24886 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — theanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (L-theanine QD) (Experimental): Patients receive L-theanine PO QD for 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: Survey Administration; Drug: Theanine
- Arm II (L-theanine BID) (Experimental): Patients receive L-theanine PO BID for 6 weeks in the absence of unacceptable toxicity.
  Interventions: Other: Survey Administration; Drug: Theanine

INTERVENTIONS:
Other: Survey Administration — Ancillary studies
Drug: Theanine — Given L-theanine PO
  Other Names: L-theanine; N-Ethyl-L-Glutamine; Suntheanine; Theanin

SUMMARY:
This clinical trial tests the feasibility, best dose, and effectiveness of L-theanine for supporting relaxation and mood among cancer patients in surveillance. L-theanine is a substance found in the leaves of green tea with potential to enhance mental health and well-being. It works by increasing certain chemicals within the body that have been associated with stress reduction, mood stabilization, and improved cognitive performance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of L-theanine use among cancer patients in surveillance based on adherence.

II. To determine the relationship of L-theanine on relaxation and supporting mood among cancer patients in surveillance with a dose of 200mg once daily versus (vs) twice daily, as measured by Visual Analog Scale-Relaxation (VAS-R).

SECONDARY OBJECTIVES:

I. To observe the relationship of L-theanine in reducing anxiety among cancer patients in surveillance, as measured by Visual Analog Scale-Anxiety (VAS-A).

II. To observe the relationship of L-theanine on mood states as measured by Short Form of the Profile of Mood States (POMS-SF).

EXPLORATORY OBJECTIVES:

I. To determine the feasibility of L-theanine use among cancer patients in surveillance based on recruitment.

II. To observe the relationship of L-theanine in supporting sleep among cancer patients in surveillance as measured by the Pittsburgh Sleep Quality Index (PSQI).

III. To describe the side effects of L-theanine supplementation. IV. To observe the relationship between L-theanine on symptom burden among cancer patients in surveillance as measured by Edmonton Symptom Assessment Scale (ESAS).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive L-theanine orally (PO) once daily (QD) for 6 weeks in the absence of unacceptable toxicity.

ARM II: Patients receive L-theanine PO twice daily (BID) for 6 weeks in the absence of unacceptable toxicity.

After completion of study intervention, patients are followed up at 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Willingness to comply with all study interventions including the use of L-theanine and follow-up assessments
* Age: ≥ 18 years
* Ability to read and understand English or Spanish for questionnaires
* Patients must be a cancer patient who has completed treatment and has been in surveillance for at least 6 months
* Participants must not have used any herbs or supplements in the past 30 days
* Participants must report an anxiety score of > 3 on Visual Analog Scale - Anxiety
* Participants must not have had any changes to their psychiatric medications within the past 60 days
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 month after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Concurrent use of other alternative medicines, including herbal agents and high-dose vitamins and minerals, unless taken to correct a documented vitamin or mineral insufficiency
* Chemotherapy, radiation therapy, biological therapy, immunotherapy, or any other systemic treatment excluding hormonal therapy (must be on a stable dose of hormonal therapy for at least 60 days)
* Any patients taking bortezomib, as L-theanine can decrease effectiveness
* Any patients currently enrolled in other clinical trials that might interfere with the results of this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Any patients with an ongoing active/unstable psychiatric condition, depressive/bi-polar related disorders, anxiety, psychosis disorders, or substance use that may interfere with the ability to participate in the study as outlined in the study procedures section of the protocol
* Any patients with chronically unstable blood pressure or chronic low blood pressure
* Diagnosis of Gilbert's disease
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Adherence rates | Up to 8 weeks
  Will consider the study feasible if at least 75% of enrolled participants adhere to the planned intervention. Adherence will be defined as having at least 75% study drug accountability. Will be estimated along with the 95% exact binomial confidence interval.
Perceived levels of relaxation | From baseline to day 42
  Measured via Visual Analog Scale-Relaxation (VAS-R). Response is defined as a favorable change of at least 1.5 points on the VAS-R. Will be estimated along with the 95% exact binomial confidence interval. Within-group mean changes in VAS-R will be examined using paired t-tests (comparing any two time points of interest).

SECONDARY OUTCOMES:
Self-perceived anxiety | From screening to day 42
  Assessed via Visual Analog Scale-Anxiety. Within-group mean changes will be examined using paired t-tests (comparing any two time points of interest). Between-group mean changes will be evaluated at each time point using independent-samples t-tests.
Anxiety and depression | From baseline to day 42
  Assessed via Hospital Anxiety and Depression Scale. Within-group mean changes will be examined using paired t-tests (comparing any two time points of interest). Between-group mean changes will be evaluated at each time point using independent-samples t-tests.
Transient mood states | From baseline to day 42
  Assessed via Short Form of the Profile of Mood States that includes tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment. Within-group mean changes will be examined using paired t-tests (comparing any two time points of interest). Between-group mean changes will be evaluated at each time point using independent-samples t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Veguilla, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope at Irvine Sand Canyon, Irvine, California